CLINICAL TRIAL: NCT01860677
Title: The Effects of Cranial Electrotherapy Stimulation (CES) on Brain Function, Brain Chemistry and Mood: An fMRI/MRS Study
Brief Title: The Effects of Cranial Electrotherapy Stimulation (CES) on Brain Function, Brain Chemistry and Mood
Acronym: CES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Mending Minds Foundation (Unknown)
Responsible Party: Principal Investigator, Scott Lukas, Director, McLean Imaging Center, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P-001567
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Mood
Keywords: cranial stimulation; BOLD (Blood Oxygenation Level Dependent); fMRI (Functional Magnetic Resonance Imaging); spectroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active stimulation (Active Comparator): The Fisher Wallace Cranial Stimulator device generates micro currents of electricity using a patented series of radio frequencies. The device has been designated by the FDA to be minimally invasive and has FDA approval to be used to reduce symptoms associated with anxiety, depression, pain and insomnia. The unit is locked at the factory to deliver a maximal output of 4 mA of current and has a timer that prevents it from staying on longer than 20 minutes. Current will be limited to a maximum of 2 mA.
  Interventions: Device: Fisher Wallace Cranial Stimulator
- Sham stimulation (Placebo Comparator): Participants are outfitted with a device that is identical to the Fisher Wallace Cranial Stimulator in appearance but does not deliver any current.
  Interventions: Device: Fisher Wallace Cranial Stimulator

INTERVENTIONS:
Device: Fisher Wallace Cranial Stimulator — The Fisher Wallace Cranial Stimulator device generates micro currents of electricity using a patented series of radio frequencies.

SUMMARY:
Document whether the Fischer Wallace Cranial Stimulator produces any measurable changes in brain activity.

DETAILED DESCRIPTION:
The advent of an appreciation that alternative and complementary practices can have some beneficial effect on health has prompted the question of whether there are empirical measures of improvement that do not rely solely on subjective reports. The present study proposes to explore whether transcranial stimulation (or cranial electrotherapy stimulation; CES) using an FDA-approved device can alter brain function, mood and responses to cognitive tasks.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 55 years old
* Otherwise physically healthy (normal physical exam, ECG, blood and urine chemistries)
* Female participants must use medically approved method of contraception. If barrier method is used, they must agree to using two methods simultaneously (e.g., diaphragm and condom).
* If on antidepressant or antianxiety medication, must be on a stable prescription regimen with no intentions to change drugs or dose during the next 11 weeks.

Exclusion Criteria:

* Opiate maintenance (e.g., methadone or buprenorphine)
* Drug use (other than nicotine, alcohol, or marihuana) greater than 50 lifetime uses.
* Meets criteria for current drug abuse or dependence (other than nicotine, alcohol, or marihuana). Past abuse/dependence (greater than 3 years) is acceptable.
* Meets criteria for alcohol dependence. Past abuse/dependence (greater than 3 years) is acceptable. They may meet criteria for alcohol abuse.
* Physical health problems
* History of significant cardiac problems
* History of seizures
* Pregnancy
* Persons with a demand-type cardiac pacemaker
* Persons receiving vagus nerve simulation
* Persons receiving deep brain stimulation
* Participants cannot have any conditions that are contraindicated for MRI

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Lukas, PhD, Principal Investigator — McLean Imaging Center, McLean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilula MF, Barach PR. Cranial electrotherapy stimulation: a safe neuromedical treatment for anxiety, depression, or insomnia. South Med J. 2004 Dec;97(12):1269-70. doi: 10.1097/01.SMJ.0000136304.33212.06. No abstract available. PMID 15646771
- [Background] Smith RB (2006) Cranial electrotherapy stimulation: Its first fifty years, plus three: a monograph. Oklahoma: Tate Publishing & Enterprises

RESULTS

PARTICIPANT FLOW:
Groups:
- Active First, Then Sham: Active treatment first, then Sham
  Active:
  The Fisher Wallace Cranial Electrostimulation device generates micro currents of electricity using a patented series of radio frequencies. The device has been designated by the FDA to be minimally invasive and has FDA approval to be used to reduce symptoms associated with anxiety, depression, pain and insomnia. The unit is locked at the factory to deliver a maximal output of 4 mA of current and has a timer that prevents it from staying on longer than 20 minutes. Current will be limited to a maximum of 2 mA.
  Fisher Wallace Cranial Stimulator
  Sham:
  Participants are outfitted with a device that is identical to the Fisher Wallace Cranial Stimulator in appearance but does not deliver any current.
  Fisher Wallace Cranial Stimulator: The Fisher Wallace Cranial Stimulator device generates micro currents of electricity using a patented series of radio frequencies.
- Sham First, Then Active: Sham first, then Active treatment
  Active:
  The Fisher Wallace Cranial Electrostimulation device generates micro currents of electricity using a patented series of radio frequencies. The device has been designated by the FDA to be minimally invasive and has FDA approval to be used to reduce symptoms associated with anxiety, depression, pain and insomnia. The unit is locked at the factory to deliver a maximal output of 4 mA of current and has a timer that prevents it from staying on longer than 20 minutes. Current will be limited to a maximum of 2 mA.
  Fisher Wallace Cranial Stimulator
  Sham:
  Participants are outfitted with a device that is identical to the Fisher Wallace Cranial Stimulator in appearance but does not deliver any current.
  Fisher Wallace Cranial Stimulator: The Fisher Wallace Cranial Stimulator device generates micro currents of electricity using a patented series of radio frequencies.
Period: First Intervention (1 Day)
Arm/Group | Active First, Then Sham | Sham First, Then Active
Started | 8 | 0
Completed | 8 | 0
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Active First, Then Sham | Sham First, Then Active
Started | 8 | 0
Completed | 1 | 0
Not Completed | 7 | 0
Not completed — Lost to Follow-up | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All of the study participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Caffeine consumption [Mean (Standard Deviation); unit: caffeinated beverages/week] | 5.2 (6.1)
Alcohol consumption [Mean (Standard Deviation); unit: alcoolic drinks/week] | 2.1 (2.1)
Marihuana use (spelling with 'h' used by DEA and FDA) [Mean (Standard Deviation); unit: lifetime uses] | 3.5 (6.9)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.35 (4.76)

OUTCOME MEASURES:

1. Primary Outcome: BOLD fMRI (Neural Activation Patterns/Brain Function) Among Participants Who Completed Both Active and Sham Stimulation Visits
Description: Quantitative changes in neural activation patterns during task performance as measured by BOLD functional MRI from 20 minutes of CES compared to pre-treatment.
  The coupling ratio is defined as the percent change in the cerebral blood flow divided by the percent change in the cerebral metabolic rate of oxygen consumption.
Time Frame: within 30 minutes after CES treatment concluded; pre-treatment is at least 20 minutes before end of treatment
Population: Data were not collected
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: BOLD fMRI (Neural Activation Patterns/Brain Function) in Active Stimulation Arm Only
Description: as for outcome 1
Time Frame: within 30 minutes after CES treatment concluded; pre-treatment is at least 20 minutes before end of treatment
Population: Data were not collected for Sham intervention; Outcome pre-specified to be assessed for Active Arm only
Measure: Mean (Standard Deviation); unit: coupling ratio
Groups:
- Active Stimulation: The Fisher Wallace Cranial Electrostimulation device generates micro currents of electricity using a patented series of radio frequencies. The device has been designated by the FDA to be minimally invasive and has FDA approval to be used to reduce symptoms associated with anxiety, depression, pain and insomnia. The unit is locked at the factory to deliver a maximal output of 4 mA of current and has a timer that prevents it from staying on longer than 20 minutes. Current will be limited to a maximum of 2 mA.
  Fisher Wallace Cranial Stimulator
Arm/Group | Active Stimulation
Number analyzed (Participants) | 8
coupling ratio | 0.2 (0.5)

3. Secondary Outcome: Change in Positive and Negative Affect Schedule (PANAS) in Active Stimulation Arm
Description: Positive and Negative Affect Schedule (PANAS), as defined by Watson et al. (1988), range between 10 and 50 points. Anchors of "not at all" (10) to "most ever" (50) were used to rank each measure. Change compares post-treatment to pre-treatment.
  Positive Affects included the following terms: Attentive, Active, Alert, Excited, Enthusiastic, Determined, Inspired, Proud, Interested, and Strong. Negative Affects included the following terms: Hostile, Irritable, Ashamed, Guilty, Distressed, Upset, Scared, Afraid, Jittery, and Nervous. Higher positive affect scores indicated a better outcome, while lower negative affect scores indicated a better outcome.
Time Frame: within 30 minutes after CES treatment concluded; pre-treatment is at least 20 minutes before end of treatment
Population: Participants in the active stimulation arm. Data were not collected for Sham intervention; Outcome pre-specified to be assessed for Active Arm only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Stimulation
Number analyzed (Participants) | 8
units on a scale
  PANAS Positive Affect | 1.88 (3.60)
  PANAS Negative Affect | -0.63 (0.74)

4. Secondary Outcome: Change in Visual Analogue Scale (VAS) in Active Stimulation Arm
Description: Visual Analogue Scale (VAS) ranges from 0-100. Anchors of "not at all" (0) to "most ever" (100) were used to rank the following:
  anxious, sleepy, dizzy, relaxed, physical symptoms, confused, sluggish, energetic, fatigued, and stressed. Change compares post-treatment to pre-treatment.
Time Frame: within 30 minutes after 1-day CES treatment concluded; pre-treatment is at least 20 minutes before end of treatment
Population: Data were not collected for Sham intervention; Outcome pre-specified to be assessed for Active Arm only.
  3 participants were missing data on these measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Stimulation
Number analyzed (Participants) | 5
units on a scale
  Anxiety | -2.90 (5.85)
  Sleepy | 5.80 (21.06)
  Dizzy | 1.10 (6.42)
  Relaxed | -2.60 (12.77)
  Physical symptoms | 2.30 (2.71)
  Confused | 0.80 (1.89)
  Sluggish | -1.80 (18.70)
  Energetic | 0.00 (9.56)
  Fatigued | 3.80 (6.52)
  Stressed | -3.40 (5.67)

ADVERSE EVENTS:
Description: Only one participant completed the Sham intervention.
Groups:
- Sham Stimulation: Participants are outfitted with a device that is identical in appearance but does not deliver any current.
Arm/Group | Active Stimulation | Sham Stimulation
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/1
Other Adverse Events (participants affected / at risk) | 0/8 | 0/1

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No